CLINICAL TRIAL: NCT00597636
Title: Genetic Susceptibility to Lung Cancer in Never Smokers
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 05-038
Record Dates: First submitted 2008-01-10; First posted 2008-01-18 (Estimated); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Lung Cancer
Keywords: smokers
MeSH Terms: conditions — Lung Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood

GROUPS / COHORTS (2):
- 1: NEVER SMOKERS WITH LUNG CANCER
  Interventions: Behavioral: Questionaire, blood sample
- 2: NEVER SMOKERS WITHOUT ANY CANCER
  Interventions: Behavioral: Questionaire, Blood sample

INTERVENTIONS:
Behavioral: Questionaire, blood sample — Provide 30ml blood for laboratory assays Complete Health Questionnaire
  Groups: 1
Behavioral: Questionaire, Blood sample — Provide 30ml blood for laboratory assays Complete Health Questionnaire
  Groups: 2

SUMMARY:
The purpose of this study is to help us better understand the cellular changes that may lead to the development of lung cancer. We want to compare people who have never smoked and yet have been diagnosed with lung cancer to never smokers who have not developed lung cancer. We hope to use the information obtained in this study as the basis for future studies and will not regard the results from this study as final.

ELIGIBILITY:
Inclusion Criteria:

* Cases will be eligible for inclusion if:
* They have been diagnosed with a lung cancer or have had previous surgical treatment for their lung cancer and have smoked fewer than 100 cigarettes in their lifetime, are/were not regular cigar or pipe smokers, and
* They have had no prior chemotherapy or radiation treatment within the last year (Exception: genotyping analysis/screening can be performed on specimens from individuals who had chemo/radiation treatment within the last year as germline DNA will not be affected)
* They speak and read English
* They understand and agree to sign informed consent, and
* They agree to give us a blood sample, and
* They agree to complete the study questionnaire, and
* They agree to have their pathology information reviewed by study personnel.
* Controls will be eligible for inclusion if:
* They have not been diagnosed with any type of cancer, exclusive of nonmelanoma skin cancer and have smoked fewer than 100 cigarettes in their lifetime, are/were not regular cigar or pipe smokers, and
* They speak and read English
* They understand and agree to sign informed consent, and
* They agree to give us a blood sample, and
* They agree to complete the study questionnaire.

Exclusion Criteria:

* Subjects who do not meet the inclusion criteria for either the case or control groups will not be eligible for this study.
* All individuals who otherwise meet the eligibility requirements above, but who have had chemotherapy or radiation therapy within 1 year of evaluation will be excluded (Exception: genotyping analysis/screening can be performed on specimens from individuals who had chemo/radiation treatment within the last year as germline DNA will not be affected).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: MSKCC clinics
Sampling Method: Non-Probability Sample
Enrollment: 238 (Actual)
Dates: Start 2005-06; Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
To evaluate germline genetic variants and their association with lung cancer in never smokers. | conclusion of study

SECONDARY OUTCOMES:
To evaluate whether overall DNA damage/repair capacity is associated with lung cancer in never smokers. | conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: Irene Orlow, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org